CLINICAL TRIAL: NCT00671957
Title: Energy Expenditure and Gastric Bypass Surgery Study
Acronym: Energy
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bruce Wolfe, Professor of Surgery, Oregon Health and Science University
Other Study IDs: IRB00002212
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Morbid Obesity
Keywords: Obesity; Bariatric; Surgery; Activity
MeSH Terms: conditions — Obesity, Morbid; Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing gastric bypass: Patients undergoing gastric bypass surgery and who are participants in Longitudinal Assessment of Bariatric Surgery (LABS-2).
  Inclusion Criteria:
  * No acute illnesses
  * Weight less than 227 kg (limit of Bod Pod and Treadmill)
  * Able to walk at 2.4 mph for 15 minutes (needed for the energy expenditure testing)
  * No tobacco use
  * Ability to stop alcohol consumption during test phases
  * For female subjects; no plans for pregnancy in 24 months and menstrual cycles of 21-35 days
  * No history of eating disorder
  * No history of current substance abuse
  * No history of chest pain or shortness of breath at rest or on exertion.
  * Negative pregnancy in women.

SUMMARY:
The aim of this study is to assess whether the energy you burn daily increases after you have bariatric surgery. Until now, there hasn't been an effective way of measuring all activity on a daily basis. Physical Activity Monitoring System (PAMS) has been created just for this purpose. PAMS is a garment that can be worn under your clothes, that records body position and movement through space. We will use the PAMS along with special water to measure your total daily energy expenditure right before surgery, and again 6 months and 24 months after surgery.

Study subjects will be initially recruited from OHSU IRB-Approved advertisements. Interested study subjects will be screened through an informal telephone interview. If there are no health conditions that exclude participation, subjects will be asked to give IRB-approved consent.

Subjects will be consenting to undergo three 18 day phases. Each phase will consist of 15 daily visits to the Clinical & Translational Research Center (CTRC), and 3 full day and nights in the CTRC.

DETAILED DESCRIPTION:
The aim of this study is to assess whether the energy you burn daily increases after you have bariatric surgery. Until now, there hasn't been an effective way of measuring all activity on a daily basis. Physical Activity Monitoring System (PAMS) has been created just for this purpose. PAMS is a garment that can be worn under your clothes, that records body position and movement through space. We will use the PAMS along with special water to measure your total daily energy expenditure right before surgery, and again 6 months and 24 months after surgery.

Study subjects will be initially recruited from OHSU IRB-Approved advertisements. Interested study subjects will be screened through an informal telephone interview. If there are no health conditions that exclude participation, subjects will be asked to give IRB-approved consent.

Subjects will be consenting to undergo three 18 day phases. Each phase will consist of 15 daily visits to the Clinical & Translational Research Center (CTRC), and 3 full day and nights in the CTRC. The CTRC day visits will be 1 hour visits, where subjects will shower, replace their dirty PAMS with a clean PAMS, have their weight measured and be asked to walk on a treadmill for a total of 12 minutes with 3 minutes each at 0.0, 0.6, 1.6 and 2.4 mph. Subjects will be asked to drink special water on Day 2, and daily urine samples will be collected for 14 days. On Day 16 subjects will undergo a series of Energy Expenditure tests using a breath analyzer. Subjects will begin with lying for 30 minutes, then sitting for 20 minutes, standing for 20 minutes, and a transitional period of standing and sitting for 20 minutes. Subjects will then be asked to walk for three 15 minute intervals at 0.8, 1.6, and 2.4 mph. Day 17 will be a repeat of Day 16 but will be followed by Dual Energy X-Ray Absorptiometry (DEXA) or BodPod (for individuals over 350 lbs) which is device which uses the movement of air to measure your muscle and fat volumes. Day 18 subjects will begin with lying for 30 minutes,then be given a breakfast to eat. Their breathing test will then continue every 15 of 30 minutes after eating breakfast to assess how much energy their body burns during digestion, for 450 minutes (7.5 hours).

PAMS allows physical activity to be measured precisely during daily activities. By attaching sensors (inclinometers) to the torso and thigh, body posture can be defined:

Lying: torso and thigh sensors indicate horizontal, Standing: torso and thigh sensors indicate vertical, Sitting: torso sensor = vertical, thigh sensor = horizontal. Duplicate sensor sets are used in all subjects to gather duplicate data every ½ second for 14 days. The physical activity data are combined with the breath measurement data to allow us to measure all forms of activity. The following are key features; specialized sensors (accelerometers) are completely integrated with the inclinometers so that data on body position and movement are continuously gathered; the sensors are attached to the subject using a harnesses that allows a full range of daytime and nighttime physical activities as well as bathroom use.

Data analysis is simple requiring a standard PC that runs Excel and written macros programs. Once this data is downloaded, it will be sent to Mayo Rochester where it will be analyzed for the following:

* Time-spent lying, sitting, standing and walking,
* Average accelerometer output for non-walking activities (lying, sitting and standing).
* Average accelerometer output for walking and,
* Number of transitions made between postures (e.g. 'sitting-to-standing'). Breathing feedback will be used to calculate, in duplicate measurements of the Energy Expenditure (EE) of sitting, standing, transitions and walking at 0.8, 1.6 and 2.4 mph.

Posture and activity EE data collection. For the physical activity monitoring period (Days 2-15), the EE for sitting, standing and transitions will be calculated by multiplying the time engaged in each activity (or number of transitions) by the EE for that activity.

Non-Exercise Activity EE = EE sitting + EE standing + EE transitions + EE walking.

The special water will be measured in the urine collected daily. The daily urine samples will be shipped to and analyzed by University of Wisconsin's special instrument in Dr. Schoeller's lab. This special water has the ability to tell us your total energy expenditure over the whole day. The special water has a marker or label attached to the water molecule. The special instrument reads how many water molecules possess this special label. Body water excreted through urine can tell us a person's total daily energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

* No acute illnesses
* Weight less than 227 kg (limit of Bod Pod and Treadmill)
* Able to walk at 2.4 mph for 15 minutes (needed for the energy expenditure testing)
* No tobacco use
* Ability to stop alcohol consumption during test phases
* For female subjects; no plans for pregnancy in 24 months and menstrual cycles of 21-35 days
* No history of eating disorder
* No history of current substance abuse
* No history of chest pain or shortness of breath at rest or on exertion.
* Negative pregnancy in women.

Exclusion Criteria:

* Informed consent not obtained
* Prior bariatric surgery
* Unlikely to comply with follow-up protocol (e.g., travel time from home too long to make visits feasible, unwilling to return for follow-up visits)
* Unable to communicate with local study staff
* Lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbidly obese patients undergoing Bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2006-02; Primary Completion 2007-07 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
To compare physical activity and activity thermogenesis in patients undergoing gastric bypass bariatric surgery at baseline (pre-operatively) and 6 and 24 months after gastric bypass surgery. | 24 months
  To compare physical activity and activity thermogenesis in patients undergoing gastric bypass bariatric surgery at baseline (pre-operatively) and 6 and 24 months after gastric bypass surgery.

SECONDARY OUTCOMES:
To evaluate whether changes in weight correlate with changes in activity thermogenesis in patients undergoing gastric bypass surgery at baseline (pre-operatively) and 6 and 24 months after gastric bypass surgery. | 24 months
  To evaluate whether changes in weight correlate with changes in activity thermogenesis in patients undergoing gastric bypass surgery at baseline (pre-operatively) and 6 and 24 months after gastric bypass surgery.
To evaluate the changes in basal metabolic rate (BMR) and thermic effect of food (TEF) in patients undergoing gastric bypass surgery at baseline (pre-operatively) and 6 and 24 months after gastric bypass surgery. | 24 months
  To evaluate the changes in basal metabolic rate (BMR) and thermic effect of food (TEF) in patients undergoing gastric bypass surgery at baseline (pre-operatively) and 6 and 24 months after gastric bypass surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce M Wolfe, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States